CLINICAL TRIAL: NCT01567072
Title: Non Steroidal Antiinflammatory Drugs Influence on Heal of Distal Radius Fracture
Acronym: CHIP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Marius Aliuskevicius (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor-Investigator, Marius Aliuskevicius, Principal Investigator, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010-018543-34
Record Dates: First submitted 2012-03-20; First posted 2012-03-30 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Forearm Fracture
Keywords: NSAID; bone fracture; heal
MeSH Terms: conditions — Fractures, Bone | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NSAIDs in 7 days (Experimental): NSAIDs (Ibuprofen) in 7 days
  Interventions: Drug: Ibuprofen
- NSAIDs in 3 days (Active Comparator): NSAIDs (Ibuprofen) in the first 3 days and placebo in the last 4 days
  Interventions: Drug: Ibuprofen
- Placebo (Placebo Comparator): Only placebo in 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen — Treatment with Ibuprofen 600mg 3times a day in 7 days after Colles fracture diagnosis
  Other Names: M01AE01 7 days
  Arms: NSAIDs in 7 days
Drug: Ibuprofen — Treatment with Ibuprofen 600mg 3 times daily in 3 days after´diagnosis - Colles fracture
  Other Names: M01AE01 3 days
  Arms: NSAIDs in 3 days
Drug: Placebo — Only placebo treatment instead of NSAID painkillers
  Other Names: M01AE01 0 days
  Arms: Placebo

SUMMARY:
It is believed, that Non Steroidal Antiinflammatory Drug (NSAID) drugs slows bone healing, but the knowledge is based only on animal studies, and the results are automatically raised for the people.

Many patients with bone fracture must therefore avoid the formerly so popular and good painkillers, although no clinical trial evidence is, that this medicine is really harmful for patients with fractures.

The purpose of this study is to investigate whether these drugs slows bone healing, and what the relationship is between various bone studies - DEXA scanning, biochemical bone marker tests, radiographic controls and tissue examination of newly formed bone under a microscope. How sensitive and specific, each of the above study methods? If they are just as sensitive, the cheapest of them recommended as a routine investigation on suspicion of bone effects. Furthermore, to compare the benefit (pain-relieving effect, influence on rehabilitation) of these drugs and their possible harmful side effects (affected and delayed bone healing).

The expectation is that the study may contribute to increased knowledge about NSAIDs effect do pain management, rehabilitation and the entire treatment process significantly easier and safer, so that patients recover faster and return to usual activities.

ELIGIBILITY:
Inclusion Criteria:

* written acceptance to participate in the study
* immobilisation or reposition or surgery demanding Colles fracture (which needs to be fixed with external fixation).

Exclusion Criteria:

* age - younger than 50 years or older than 80 years
* treatment with prednisolon
* NSAIDs - treatment
* previous fracture or surgery at the wrist
* lack of mental and physical capacity to follow studies' instructions
* lack of informed consent
* other diseases can affect bone substance (oncology, endocrine diseases)
* medical contraindications to NSAIDs use
* smoking, alcohol consumption of more than 14 drinks per week
* secondary dislocation of fracture also apply as exclusion criterion.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2012-04; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of changes of fractures position by X rays investigation | 1 week, 2 weeks, 6 weeks
  Measurement of possible secondary dislocation

SECONDARY OUTCOMES:
DEXA - scanning | 12 weeks
  Evaluation of bone density
Bone Biochemical markers | 1 week, 2 weeks, 5 weeks, 3 months, 1 year
  Se CrossLaps ELISA, N/Mid Osteocalcin Elisa
Histomorfometrical evaluation of bone biopsy from callus area | 6 weeks
  qualitative evaluation of bone ossification

OTHER OUTCOMES:
Repeated measurements of pain in 14 days | 2 weeks
  subjective pain registration in 10 points scala 3 times dayly in 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Marius Aliuskevicius, Physician, Principal Investigator — Aalborg University Hospital
Locations (1):
- Department of Orthopaedic Surgery, Aalborg University Hospital, Aalborg, Denmark

REFERENCES:
- [Background] Persson PE, Nilsson OS, Berggren AM. Do non-steroidal anti-inflammatory drugs cause endoprosthetic loosening? A 10-year follow-up of a randomized trial on ibuprofen for prevention of heterotopic ossification after hip arthroplasty. Acta Orthop. 2005 Dec;76(6):735-40. doi: 10.1080/17453670510045309. PMID 16470423